CLINICAL TRIAL: NCT00411658
Title: Devitalized Non-valved Pulmonary Artery Allograft Implant for the Repair of Congenital Cardiac Abnormalities
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Submission converted to 510(k)
Sponsor: LifeNet Health (Industry)
Other Study IDs: CR06-002
Record Dates: First submitted 2006-12-13; First posted 2006-12-14 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: NA-Study Withdrawn
MeSH Terms: interventions — Cryopreservation

ARMS (2):
- Investigational Device (Experimental)
  Interventions: Device: Investigational Device; Device: Experimental
- Cryopreserved (Active Comparator)
  Interventions: Other: Cryopreserved

INTERVENTIONS:
Device: Investigational Device
  Arms: Investigational Device
Device: Experimental
  Arms: Investigational Device
Other: Cryopreserved
  Arms: Cryopreserved

SUMMARY:
Study no longer required

Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)